CLINICAL TRIAL: NCT04168268
Title: Influence of Post-anesthesia Care Unit Delirium After Radical Prostatectomy on Self-reported Cognitive Function and Health-related Quality of Life
Brief Title: Patient-reported Outcome Measures After Post-anesthesia Care Unit Delirium
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PACU-DE
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Delirium; Neurocognitive Disorders
MeSH Terms: conditions — Delirium; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess self-reported cognitive function and health-related quality of life in patients with and without early postoperative delirium

DETAILED DESCRIPTION:
Neurocognitive disorders including postoperative delirium are a serious complication after surgery and anesthesia in the elderly. Postoperative delirium is an acute-onset diffuse brain dysfunction that is characterized by a fluctuating course of confusion, disorganized thinking, inattention, irritability, disturbances of the circadian rhythm, and disorders of consciousness. Post-anesthesia care unit (PACU) delirium occurs immediately after emergence from anesthesia and affects up to 45% of patients after elective surgery.

It is unclear, whether PACU delirium is associated with intermediated or long-term adverse outcomes including neurocognitive disorders or mortality. The aim of this prospective observational was to assess self-reported cognitive function and health-related quality of life in patients with and without PACU delirium three months after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* elective radical prostatectomy
* >60 years
* fluent in German

Exclusion Criteria:

* preexisting cognitive impairment
* cerebrovascular disease

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective radical prostatectomy for prostate cancer at a high-volume prostate cancer center were screened on the day before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Self-reported cognitive failures | three months
  Cognitive Failures Questionnaire

SECONDARY OUTCOMES:
Health-related quality of life | three months
  Short Form Health Survey 36

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kainz E, Stuff K, Kahl U, Wiessner C, Yu Y, von Breunig F, Nitzschke R, Haese A, Graefen M, Fischer M. Impact of postanesthesia care unit delirium on self-reported cognitive function and perceived health status: a prospective observational cohort study. Qual Life Res. 2022 Aug;31(8):2397-2410. doi: 10.1007/s11136-022-03087-1. Epub 2022 Jan 27. PMID 35084649